CLINICAL TRIAL: NCT03217747
Title: Phase I/II Study to Evaluate the Safety and Tolerability of Avelumab in Combination With Other Anti-Cancer Therapies in Patients With Advanced Malignancies
Brief Title: Avelumab, Utomilumab, Anti-OX40 Antibody PF-04518600, and Radiation Therapy in Treating Patients With Advanced Malignancies
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-0014; NCI-2018-01118 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2017-0014 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2017-07-12; First posted 2017-07-14 (Actual); Results first posted 2025-10-14 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Advanced Malignant Solid Neoplasm; Castration-Resistant Prostate Carcinoma; Malignant Solid Neoplasm; Metastatic Malignant Solid Neoplasm; Metastatic Prostate Carcinoma; Prostate Carcinoma Metastatic in the Bone; Refractory Malignant Solid Neoplasm; Stage IV Prostate Cancer AJCC v8; Stage IVA Prostate Cancer AJCC v8; Stage IVB Prostate Cancer AJCC v8
MeSH Terms: conditions — Neoplasm Metastasis; Prostatic Neoplasms | interventions — avelumab; Radiotherapy; Radiation; utomilumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Arm A (utomilumab, avelumab) (Experimental): Patients receive utomilumab IV over 60 minutes on day 1 of each cycle and avelumab IV over 60 minutes on days 1 and 15 beginning day 15 of cycle 1. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Avelumab; Biological: Utomilumab
- Arm B (PF-04518600, avelumab) (Experimental): Patients receive anti-OX40 agonist monoclonal antibody PF-04518600 IV over 60 minutes on days 1 and 15 of each cycle and avelumab IV over 60 minutes on days 1 and 15 beginning day 15 of cycle 1. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Avelumab; Biological: Ivuxolimab
- Arm C (PF-04518600, utomilumab, avelumab) (Experimental): Patients receive anti-OX40 agonist monoclonal antibody PF-04518600 IV over 60 minutes on days 1 and 15 of each cycle, utomilumab over 60 minutes on day 1, and avelumab IV over 60 minutes on days 1 and 15 beginning day 15 of cycle 1. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Avelumab; Biological: Ivuxolimab; Biological: Utomilumab
- Arm D (avelumab, utomilumab, radiation therapy) (Experimental): Patients undergo radiation therapy on days -5 to -1. Patients receive avelumab IV over 60 minutes on days 1 and 15 of beginning day 15 of cycle 1 and utomilumab IV over 60 minutes on day 1. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Avelumab; Radiation: Radiation Therapy; Biological: Utomilumab
- Arm E (avelumab, PF-04518600, radiation therapy) (Experimental): DISCONTINUED AS OF AMENDMENT 9 (02/11/2020) Patients undergo radiation therapy on days -14 to -1. Patients receive avelumab IV over 60 minutes on days 1 and 15 beginning day 15 of cycle 1 and anti-OX40 agonist monoclonal antibody PF-04518600 IV over 60 minutes on days 1 and 15, and. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Avelumab; Biological: Ivuxolimab; Radiation: Radiation Therapy
- Arm F (avelumab, PF-04518600, radiation therapy) (Experimental): DISCONTINUED AS OF AMENDMENT 9 (02/11/2020) Patients undergo radiation therapy on days -14 to -1. Patients receive avelumab IV over 60 minutes on days 1 and 15 beginning day 15 of cycle 1, utomilumab IV over 60 minutes on day 1, and anti-OX40 agonist monoclonal antibody PF-04518600 IV on days 1 and 15. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Avelumab; Biological: Ivuxolimab; Radiation: Radiation Therapy; Biological: Utomilumab

INTERVENTIONS:
Drug: Avelumab — Given IV
  Other Names: Bavencio; MSB-0010718C; MSB0010718C
Biological: Ivuxolimab — Given IV
  Other Names: Anti-OX40 Agonist Monoclonal Antibody PF-04518600; PF-04518600; PF-8600; PF04518600
  Arms: Arm B (PF-04518600, avelumab); Arm C (PF-04518600, utomilumab, avelumab); Arm E (avelumab, PF-04518600, radiation therapy); Arm F (avelumab, PF-04518600, radiation therapy)
Radiation: Radiation Therapy — Undergo radiation therapy
  Other Names: Cancer Radiotherapy; ENERGY_TYPE; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation
  Arms: Arm D (avelumab, utomilumab, radiation therapy); Arm E (avelumab, PF-04518600, radiation therapy); Arm F (avelumab, PF-04518600, radiation therapy)
Biological: Utomilumab — Given IV
  Other Names: PF 05082566; PF 5082566; PF-05082566; PF-2566
  Arms: Arm A (utomilumab, avelumab); Arm C (PF-04518600, utomilumab, avelumab); Arm D (avelumab, utomilumab, radiation therapy); Arm F (avelumab, PF-04518600, radiation therapy)

SUMMARY:
This phase I/II trial studies the side effects of avelumab when given in different combinations with utomilumab, anti-OX40 antibody PF-04518600, and radiation therapy in treating patients with malignancies that have spread to other places in the body (advanced). Immunotherapy with monoclonal antibodies, such as avelumab, utomilumab, and anti-OX40 antibody PF-04518600, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Radiation therapy uses high-energy rays to kill tumor cells and shrink tumors. It is not yet known how well avelumab works in combination with these other anti-cancer therapies in patients with advanced malignancies.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. For Arm D, to establish the safety, tolerability, and dose-limiting toxicities (DLTs) of different treatment combinations of avelumab when administered in combination with a checkpoint agonist with radiation in patients with metastatic solid tumors in order to estimate the maximum tolerated dose (MTD) and select the recommended phase 2 dose (RP2D).

II. To correlate pre- and post-treatment CD8 expression with clinical benefit (complete response [CR], partial response [PR], or stable disease [SD] for > 6 months).

SECONDARY OBJECTIVES:

I. To evaluate the efficacy of the different treatment combinations in patients with metastatic solid tumors by assessing objective response rate (ORR) per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 and immune-related RECIST (irRECIST).

II. To evaluate the efficacy of the different treatment combinations in patients with metastatic solid tumors by assessing progression-free survival (PFS), duration of response (DOR), and overall survival (OS).

EXPLORATORY OBJECTIVES:

I. To understand the mechanism of action of the avelumab plus an immune modulator combination, as well as potential mechanisms of resistance.

II. To characterize the effect of avelumab combinations on immune biomarkers in peripheral blood and tumor tissue obtained from subjects pre- and post-treatment.

III. To compare the response in irradiated versus non-irradiated lesions in Arm D.

IV. To investigate immune biomarkers that are potentially predictive of response and resistance with the combination of avelumab and an immune modulator.

OUTLINE: Patients are assigned to 1 of 6 arms.

ARM A: Patients receive utomilumab intravenously (IV) over 60 minutes on day 1 of each cycle and avelumab IV over 60 minutes on days 1 and 15 beginning day 15 of cycle 1. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

ARM B: Patients receive anti-OX40 agonist monoclonal antibody PF-04518600 IV over 60 minutes on days 1 and 15 of each cycle and avelumab IV over 60 minutes on days 1 and 15 beginning day 15 of cycle 1. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

ARM C: Patients receive anti-OX40 agonist monoclonal antibody PF-04518600 IV over 60 minutes on days 1 and 15 of each cycle, utomilumab over 60 minutes on day 1, and avelumab IV over 60 minutes on days 1 and 15 beginning day 15 of cycle 1. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

ARM D: Patients undergo radiation therapy on days -5 to -1. Patients receive avelumab IV over 60 minutes on days 1 and 15 of beginning day 15 of cycle 1 and utomilumab IV over 60 minutes on day 1. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

ARM E: DISCONTINUED AS OF AMENDMENT 9 (02/11/2020) Patients undergo radiation therapy on days -14 to -1. Patients receive avelumab IV over 60 minutes on days 1 and 15 beginning day 15 of cycle 1 and anti-OX40 agonist monoclonal antibody PF-04518600 IV over 60 minutes on days 1 and 15, and. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

ARM F: DISCONTINUED AS OF AMENDMENT 9 (02/11/2020) Patients undergo radiation therapy on days -14 to -1. Patients receive avelumab IV over 60 minutes on days 1 and 15 beginning day 15 of cycle 1, utomilumab IV over 60 minutes on day 1, and anti-OX40 agonist monoclonal antibody PF-04518600 IV on days 1 and 15. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients will be followed up at 30 days and then every 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be refractory to, or intolerant of, established therapy known to provide clinical benefit for their conditions, or where subjects refuse existing therapies.
* Subjects must have measurable disease (RECIST v 1.1) or patients may have bone metastatic disease evaluable by Prostate Cancer Working Group 2 (PCWG2) for subjects with metastatic castration-resistant prostate cancer (CRPC) or according to tumor evaluation criteria best suitable and accepted for the tumor type evaluated.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
* Platelets >= 100 x 10^9/L (For patients with hepatocellular carcinoma, platelets >= 70 x 10^9/L).
* Hemoglobin >= 9 g/dL.
* Absolute neutrophil count (ANC) >= 1.5 x 10^9/L.
* White blood cell (WBC) >= 3 x 10^9/L.
* Alanine transaminase (ALT) =< 2.5 x upper normal limit (ULN) (=< 5 x ULN for subjects with documented metastatic disease to the liver).
* Aspartate aminotransferase (AST) =< 2.5 x ULN (=< 5 x ULN for subjects with documented metastatic disease to the liver).
* Alkaline phosphatase < 4 x ULN.
* Total bilirubin =< 1.5 x ULN (In the expansion cohort, subjects with Gilbert's syndrome [hereditary indirect hyperbilirubinemia] who must have a total bilirubin of =< 3 x ULN).
* Albumin >= 3 g/dL.
* Serum creatinine =< 2 x upper limit of normal (ULN) or estimated creatinine clearance >= 30 ml/min as calculated using the Cockcroft-Gault formula.
* Subject has recovered to grade =< 1 by the National Cancer Institute Common Terminology Criteria for Adverse Events, version 4.03 (NCI-CTCAE v 4.03) from the effects of recent surgery, radiotherapy, chemotherapy, hormonal therapy, or other targeted therapies, with the exception of alopecia. The exceptions for such effects are allowed lab values of =< grade 2 specified elsewhere in these inclusion criteria.
* Life expectancy of at least 12 weeks.
* Negative serum pregnancy test in women of childbearing potential within 7 days of first dose of treatment and patients of child-bearing potential must agree to use effective contraception during and after 90 days post dose. A woman of childbearing potential is defined as a premenopausal female capable of becoming pregnant. This includes women on oral, injectable or mechanical contraception; women who are single and women whose male sexual partners have been vasectomized or whose male sexual partners have received or are utilizing mechanical contraceptive devices.
* Subjects must have biopsiable disease. For Arms A, B, and C, subjects must have at least two lesions amenable to biopsy and response evaluation. For Arm D subjects should have at least three lesions amenable to biopsy, response evaluation, and radiation. Tumor lesions used for biopsy should not be lesions used as RECIST target lesions. However, if patients in Arm D do not have three separate lesions, patients will be eligible if there are two lesions, in which one is > 2 centimeters (short axis) and can be used for both biopsy and response evaluation.
* Subjects must give informed consent according to the rules and regulations of the individual participating sites.

Exclusion Criteria:

* Subjects with primary central nervous system (CNS) tumor or CNS tumor involvement. However, subjects with metastatic CNS tumors may participate in this study if the subject is:

  * > 4 weeks from prior therapy completion (including radiation and/or surgery)
  * Clinically stable with respect to the CNS tumor at the time of study entry
  * Not receiving steroid therapy in treating CNS tumor or CNS tumor involvement
  * Not receiving anti-convulsive medications (that were started for brain metastases).
* Major surgery, radiation therapy or systemic anti-cancer therapy within 4 weeks of study drug administration (6 weeks for mitomycin C or nitrosoureas). Palliative radiotherapy to a limited field is allowed after consultation with the medical monitor at any time during study participation, including during screening, unless it's clearly indicative of disease progression.
* Subjects with prior anti-PD-1, anti-PD-L1 treatment. For Arms A and D, subjects may not have had prior 4-1BB treatment. For Arm B, subjects may not have had prior OX40 treatment. For Arm C, subjects may not have had prior 4-1BB or OX40 treatment.
* Diagnosis or recurrence of invasive cancer other than the present cancer within 3 years (except basal or squamous cell carcinoma of the skin that has been definitively treated).
* Clinically significant (i.e., active) cardiovascular disease: cerebral vascular accident/stroke (< 6 months prior to enrollment), myocardial infarction (< 6 months prior to enrollment), unstable angina, congestive heart failure (>= New York Heart Association classification class II), or serious cardiac arrhythmia requiring medication.
* Active infection requiring systemic therapy.
* Treatment with an investigational anti-cancer study drug within 4 weeks prior to study drug administration date.
* Concurrent therapy with approved or investigational anticancer therapeutics.
* Known prior severe hypersensitivity to investigational product(s) or any component in its formulations, including known severe hypersensitivity reactions to monoclonal antibodies (NCI CTCAE v 4.03 grade >= 3).
* Current use of immunosuppressive medication, EXCEPT for the following: a. intranasal, inhaled, topical steroids, or local steroid injection (e.g., intra-articular injection); b. systemic corticosteroids at physiologic doses =< 10 mg/day of prednisone or equivalent; c. steroids as premedication for hypersensitivity reactions (e.g., computed tomography [CT] scan premedication).
* Active autoimmune disease that might deteriorate when receiving an immuno-stimulatory agent. Patients with diabetes type I, vitiligo, psoriasis, or hypo- or hyperthyroid diseases not requiring immunosuppressive treatment are eligible.
* Prior organ transplantation including allogenic stem-cell transplantation.
* Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome.
* Hepatitis B virus (HBV) or hepatitis C virus (HCV) infection at screening (positive HBV surface antigen or HCV ribonucleic acid (RNA) if anti-HCV antibody screening test positive).
* Vaccination (live attenuated virus) within 4 weeks of the first dose of avelumab and while on trials is prohibited except for administration of inactivated vaccines.
* Persisting toxicity related to prior therapy (NCI CTCAE v. 4.03 Grade > 1); however, alopecia, sensory neuropathy grade =< 2, or other grade =< 2 not constituting a safety risk based on investigator's judgment are acceptable.
* Other severe acute or chronic medical conditions including colitis, inflammatory bowel disease, pneumonitis, pulmonary fibrosis or psychiatric conditions including recent (within the past year) or active suicidal ideation or behavior; or laboratory abnormalities that may increase the risk associated with study participation or study treatment administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study.
* Medical, psychological or social conditions that may interfere with the patient's participation in the study or evaluation of the study results.
* Pregnancy or lactation.
* Men whose partner is a woman of child-bearing potential, (i.e. biologically able to conceive), and who is not employing two forms of highly effective contraception. Highly effective contraception (e.g. male condom with spermicide, diaphragm with spermicide, intra-uterine device) must be used by both sexes during the study and must be continued for 90 days after the end of study treatment. Women of child-bearing potential is defined as sexually mature women who are not surgically sterile or who have not been naturally postmenopausal for at least 12 consecutive months (e.g., who has had menses any time in the preceding 12 consecutive months).
* A diagnosis of active scleroderma, lupus, or other rheumatologic disease which in the opinion of the treating radiation oncologist precludes safe radiation therapy.
* Has had prior radiation therapy within the past 3 months where the high dose area of the prior radiation would overlap with the high dose area of the intended radiation based on the judgement of the treatment oncologist.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 173 (Actual)
Dates: Start 2017-08-02 (Actual); Primary Completion 2025-09-02 (Actual); Study Completion 2026-04-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Aung Naing, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Lermi NO, Gouda MA, Ahmed J, Jiang X, Lee Y, Mohanty V, Derbala M, Stephen B, Jhingran A, Mohammad MM, Joo D, Francisco-Cruz A, Chen H, Calderon LA, Laberiano C, Arrechedera C, Pandurengan R, Gurses S, Yang Y, Soto LMS, Ahnert JR, Chen K, Meric-Bernstam F, Koay EJ, Javle M, Haymaker C, Naing A. Tumor microenvironment changes after treatment with avelumab and immune- stimulating agent combinations in patients with advanced solid tumors. Res Sq [Preprint]. 2026 Jan 19:rs.3.rs-7775526. doi: 10.21203/rs.3.rs-7775526/v1. PMID 41646361
- [Derived] Ahmed J, Knisely A, Torrado C, Stephen B, Yang Y, Song J, Alshawa A, Zarifa A, Jhingran A, Koay EJ, Morris VK, Javle M, Wolff RA, Meric-Bernstam F, Pant S, Rodon J, Naing A. A phase I/II trial of avelumab combinations with ivuxolimab, utomilumab, and radiation therapy in patients with advanced gastrointestinal malignancies. Oncologist. 2025 Mar 10;30(3):oyaf032. doi: 10.1093/oncolo/oyaf032. PMID 40139261

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is an open label, single center Phase I/II combination study to evaluate safety, pharmacodynamics, and anti-tumor activity of avelumab in combination with other cancer immunotherapies in Pfizer pipeline with or without radiation (XRT), in patients within metastatic cancers at The University of Texas MD Anderson Cancer Center.
Pre-assignment Details: Of the 173 patients enrolled, only 111 patients received at least 1 dose of the study agents. The remaining 62 patients screen failed and did not receive any dose of the study drugs. Per the protocol, all 111 patients who received one or more doses of drug were included in the analysis and the results are reported here.
Groups:
- Arm A Exp Avelumab Starting From C1D15; Arm A Exp Avelumab Starting From C3D1: Avelumab: 10 mg/kg IV every 2 weeks Utomilumab: 100 mg IV every 4 weeks
- Arm B Exp Avelumab Starting From C1D15: Avelumab: 10 mg/kg IV every 2 weeks Ivuxolimab: 0.3 mg/kg IV every 2 weeks Ivuxolimab: Given IV
  Utomilumab: Given IV
- Arm B Exp Avelumab Starting From C3D1: Avelumab: 10 mg/kg IV every 2 weeks Ivuxolimab: 0.3 mg/kg IV every 2 weeks
  Utomilumab: Given IV
- Arm C Escalation Avelumab Starting From C1D1: Avelumab: 10 mg/kg IV every 2 weeks Ivuxolimab: 0.3 mg/kg IV every 2 weeks Utomilumab: 20 mg IV every 4 weeks
  Ivuxolimab: Given IV
  Radiation Therapy: Undergo radiation therapy
- Arm C Exp Avelumab Starting From C1D15: Avelumab: 10 mg/kg IV every 2 weeks Ivuxolimab: 0.3 mg/kg IV every 2 weeks Utomilumab: 20 mg IV every 4 weeks
  Avelumab: Given IV
  Ivuxolimab: Given IV
  Radiation Therapy: Undergo radiation therapy
  Utomilumab: Given IV
- Arm C Exp Avelumab Starting From C3D1: Avelumab: 10 mg/kg IV every 2 weeks Ivuxolimab: 0.3 mg/kg IV every 2 weeks Utomilumab: 20 mg IV every 4 weeks
- Arm D Esc Schedule-1 Dose Level 1; XRT: Starting C1D2 to C1D11; Arm D Esc Schedule-2 Dose Level 1; XRT: Starting Days -14 to -1; Arm D Esc Schedule-3 Dose Level 1; XRT: Starting C1D1 to C1D3: Avelumab: 10 mg/kg IV every 2 weeks Utomilumab: 20 mg IV every 4 weeks XRT: 60 Gy for 10 fractions
- Arm E Esc Schedule-1 Dose Level 1; XRT: Starting C1D2 to C1D11; Arm E Esc Schedule-2 Dose Level 1; XRT: Starting Days -14 to -1: Avelumab: 10 mg/kg IV every 2 weeks Ivuxolimab: 0.3 mg/kg IV every 2 weeks XRT: 60 Gy for 10 fractions
- Arm F Esc Schedule-1 Dose Level 1; Avelumab Starting From C1D1, XRT: Starting C1D2 to C1D11; Arm F Esc Schedule-2 Dose Level 1; Avelumab Starting From C1D15, XRT: Starting Days -14 to -1: Avelumab: 10 mg/kg IV every 2 weeks Ivuxolimab: 0.3 mg/kg IV every 2 weeks Utomilumab: 20 mg IV every 4 weeks XRT: 60 Gy for 10 fractions
Period: Overall Study
Arm/Group | Arm A Exp Avelumab Starting From C1D15 | Arm A Exp Avelumab Starting From C3D1 | Arm B Exp Avelumab Starting From C1D15 | Arm B Exp Avelumab Starting From C3D1 | Arm C Escalation Avelumab Starting From C1D1 | Arm C Exp Avelumab Starting From C1D15 | Arm C Exp Avelumab Starting From C3D1 | Arm D Esc Schedule-1 Dose Level 1; XRT: Starting C1D2 to C1D11 | Arm D Esc Schedule-2 Dose Level 1; XRT: Starting Days -14 to -1 | Arm D Esc Schedule-3 Dose Level 1; XRT: Starting C1D1 to C1D3 | Arm E Esc Schedule-1 Dose Level 1; XRT: Starting C1D2 to C1D11 | Arm E Esc Schedule-2 Dose Level 1; XRT: Starting Days -14 to -1 | Arm F Esc Schedule-1 Dose Level 1; Avelumab Starting From C1D1, XRT: Starting C1D2 to C1D11 | Arm F Esc Schedule-2 Dose Level 1; Avelumab Starting From C1D15, XRT: Starting Days -14 to -1
Started | 16 | 8 | 16 | 12 | 4 | 17 | 11 | 4 | 3 | 7 | 3 | 3 | 4 | 3
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 16 | 8 | 16 | 12 | 4 | 17 | 11 | 4 | 3 | 7 | 3 | 3 | 4 | 3
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 12 | 6 | 15 | 11 | 3 | 14 | 10 | 4 | 2 | 7 | 3 | 1 | 3 | 1
Not completed — Withdrawal by Subject | 2 | 1 | 1 | 1 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Not completed — Toxicity and progression | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Removal of sole target lesion | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Stroke | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A Exp Avelumab Starting From C1D15 | Arm A Exp Avelumab Starting From C3D1 | Arm B Exp Avelumab Starting From C1D15 | Arm B Exp Avelumab Starting From C3D1 | Arm C Escalation Avelumab Starting From C1D1 | Arm C Exp Avelumab Starting From C1D15 | Arm C Exp Avelumab Starting From C3D1 | Arm D Esc Schedule-1 Dose Level 1; XRT: Starting C1D2 to C1D11 | Arm D Esc Schedule-2 Dose Level 1; XRT: Starting Days -14 to -1 | Arm D Esc Schedule-3 Dose Level 1; XRT: Starting C1D1 to C1D3 | Arm E Esc Schedule-1 Dose Level 1; XRT: Starting C1D2 to C1D11 | Arm E Esc Schedule-2 Dose Level 1; XRT: Starting Days -14 to -1 | Arm F Esc Schedule-1 Dose Level 1; Avelumab Starting From C1D1, XRT: Starting C1D2 to C1D11 | Arm F Esc Schedule-2 Dose Level 1; Avelumab Starting From C1D15, XRT: Starting Days -14 to -1 | Total
Number analyzed (Participants) | 16 | 8 | 16 | 12 | 4 | 17 | 11 | 4 | 3 | 7 | 3 | 3 | 4 | 3 | 111
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 11 | 7 | 12 | 7 | 3 | 11 | 9 | 4 | 3 | 5 | 2 | 1 | 3 | 3 | 81
  >=65 years | 5 | 1 | 4 | 5 | 1 | 6 | 2 | 0 | 0 | 2 | 1 | 2 | 1 | 0 | 30
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 8 | 11 | 11 | 1 | 12 | 3 | 4 | 2 | 5 | 1 | 2 | 2 | 1 | 72
  Male | 7 | 0 | 5 | 1 | 3 | 5 | 8 | 0 | 1 | 2 | 2 | 1 | 2 | 2 | 39
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 2 | 1 | 0 | 2 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 12
  Not Hispanic or Latino | 14 | 7 | 14 | 10 | 4 | 15 | 11 | 4 | 2 | 6 | 2 | 2 | 4 | 3 | 98
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 3 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Black or African American | 0 | 0 | 3 | 2 | 2 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 10
  White | 13 | 6 | 12 | 10 | 2 | 12 | 9 | 4 | 2 | 7 | 1 | 3 | 3 | 3 | 87
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 6
Region of Enrollment [Number; unit: participants]
  United States | 16 | 8 | 16 | 12 | 4 | 17 | 11 | 4 | 3 | 7 | 3 | 3 | 4 | 3 | 111

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose-limiting Toxicities (DLTs) (All Will be Graded According to CTCAEv4.03 Criteria)
Description: DLTs were adverse events (AEs) related to study drug in the first 2 cycles and fulfilled one of the following
  * Discontinuation due to drug and/or XRT-related toxicity before DLT period ends
  * Delay >28 days in receiving the next cycle due to drug and/or XRT-related toxicity
  * Hematologic
    * Gr4 neutropenia ≥7 days
    * Febrile neutropenia
    * Gr ≥3 thrombocytopenia associated with bleeding, or Gr 4 thrombocytopenia
    * Gr 4 anemia
  * Non-hematologic
    * Gr ≥3 nausea/vomiting or diarrhea ≥72 hours despite optimal supportive medications
    * Gr ≥3 fatigue ≥7 days
    * Gr≥2 pneumonitis ≥7 days despite corticosteroids
    * Gr≥3 rash ≥7 days despite treatment
    * Gr≥3 immune related toxicities ≥7 days despite corticosteroids
    * Any other Gr≥3 non-hematological toxicity (except for asymptomatic electrolytes abnormalities or hair loss which is not dose-limiting)
    * Gr≥3 AST, ALT, or total bilirubin elevation ≥7 days. Delay of treatment > 14 days due to non-hematologic toxicity
Time Frame: DLT was assessed during the first 2 cycles or 8 weeks (56 days) since C1D1 of treatment.
Population: All enrolled patients who received at least one dose of each study medication in the assigned treatment combination were evaluable for DLT. Patients who missed any doses during the DLT period for reasons unrelated to study drug and patients who are lost to follow-up due to reasons unrelated to treatment related AEs are not evaluable for DLT
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A Exp Avelumab Starting From C1D15 | Arm A Exp Avelumab Starting From C3D1 | Arm B Exp Avelumab Starting From C1D15 | Arm B Exp Avelumab Starting From C3D1 | Arm C Escalation Avelumab Starting From C1D1 | Arm C Exp Avelumab Starting From C1D15 | Arm C Exp Avelumab Starting From C3D1 | Arm D Esc Schedule-1 Dose Level 1; XRT: Starting C1D2 to C1D11 | Arm D Esc Schedule-2 Dose Level 1; XRT: Starting Days -14 to -1 | Arm D Esc Schedule-3 Dose Level 1; XRT: Starting C1D1 to C1D3 | Arm E Esc Schedule-1 Dose Level 1; XRT: Starting C1D2 to C1D11 | Arm E Esc Schedule-2 Dose Level 1; XRT: Starting Days -14 to -1 | Arm F Esc Schedule-1 Dose Level 1; Avelumab Starting From C1D1, XRT: Starting C1D2 to C1D11 | Arm F Esc Schedule-2 Dose Level 1; Avelumab Starting From C1D15, XRT: Starting Days -14 to -1
Number analyzed (Participants) | 16 | 8 | 16 | 12 | 4 | 17 | 11 | 4 | 3 | 7 | 3 | 3 | 4 | 3
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0

2. Secondary Outcome: Objective Response Rate Per RECIST v1.1
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) using CT, MRI,or PET-CT scan: Complete Response (CR),Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Objective Response (OR) = CR + PR.
Time Frame: At baseline and at 8-week intervals (± 7 days). Confirmatory scans were obtained 4-8 weeks following initial objective response. After 1 year of treatment scans at 12-week intervals (± 7 days), independent of cycle delays, assessed upto 3 years.
Population: All enrolled patients who were eligible, had received at least one cycle of therapy, and had baseline assessments and at least 1 on-study tumor assessment were considered evaluable for response. Patients who were treated and removed from study prior to on-study tumor assessment because of disease progression were also considered evaluable. In XRT arms, patients were considered evaluable on the study if patients received 75% of radiation dose
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A Exp Avelumab Starting From C1D15 | Arm A Exp Avelumab Starting From C3D1 | Arm B Exp Avelumab Starting From C1D15 | Arm B Exp Avelumab Starting From C3D1 | Arm C Escalation Avelumab Starting From C1D1 | Arm C Exp Avelumab Starting From C1D15 | Arm C Exp Avelumab Starting From C3D1 | Arm D Esc Schedule-1 Dose Level 1; XRT: Starting C1D2 to C1D11 | Arm D Esc Schedule-2 Dose Level 1; XRT: Starting Days -14 to -1 | Arm D Esc Schedule-3 Dose Level 1; XRT: Starting C1D1 to C1D3 | Arm E Esc Schedule-1 Dose Level 1; XRT: Starting C1D2 to C1D11 | Arm E Esc Schedule-2 Dose Level 1; XRT: Starting Days -14 to -1 | Arm F Esc Schedule-1 Dose Level 1; Avelumab Starting From C1D1, XRT: Starting C1D2 to C1D11 | Arm F Esc Schedule-2 Dose Level 1; Avelumab Starting From C1D15, XRT: Starting Days -14 to -1
Number analyzed (Participants) | 13 | 8 | 14 | 10 | 3 | 14 | 9 | 4 | 1 | 7 | 3 | 2 | 4 | 1
Participants | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Secondary Outcome: Objective Response Rate Per irRECIST
Description: Per Immune-related Response Evaluation Criteria In Solid Tumors Criteria (irRECIST) using CT, MRI,or PET-CT scan: Immune-related Complete Response (irCR),Disappearance of all target lesions; Immune-related Partial Response (irPR), >=30% decrease in the sum of the longest diameter of target and new lesions; OR = irCR + irPR.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A Exp Avelumab Starting From C1D15 | Arm A Exp Avelumab Starting From C3D1 | Arm B Exp Avelumab Starting From C1D15 | Arm B Exp Avelumab Starting From C3D1 | Arm C Escalation Avelumab Starting From C1D1 | Arm C Exp Avelumab Starting From C1D15 | Arm C Exp Avelumab Starting From C3D1 | Arm D Esc Schedule-1 Dose Level 1; XRT: Starting C1D2 to C1D11 | Arm D Esc Schedule-2 Dose Level 1; XRT: Starting Days -14 to -1 | Arm D Esc Schedule-3 Dose Level 1; XRT: Starting C1D1 to C1D3 | Arm E Esc Schedule-1 Dose Level 1; XRT: Starting C1D2 to C1D11 | Arm E Esc Schedule-2 Dose Level 1; XRT: Starting Days -14 to -1 | Arm F Esc Schedule-1 Dose Level 1; Avelumab Starting From C1D1, XRT: Starting C1D2 to C1D11 | Arm F Esc Schedule-2 Dose Level 1; Avelumab Starting From C1D15, XRT: Starting Days -14 to -1
Number analyzed (Participants) | 13 | 8 | 14 | 10 | 3 | 14 | 9 | 4 | 1 | 7 | 3 | 2 | 4 | 1
Participants | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

4. Secondary Outcome: Clinical Benefit Rate Per RECIST v1.1
Description: Per RECIST v1.0 using CT, MRI,or PET-CT scan: CR,Disappearance of all target lesions; PR, >=30% decrease in the sum of the longest diameter of target lesions; Progressive Disease (PD), Increase ≥20% of the sum of longest diameter compared with nadir (minimum 5 mm) or progression of non-target lesions or new lesion; Stable Disease (SD), Neither PR nor PD; Clinical benefit (CB) = CR + PR + SD ≥6 months.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A Exp Avelumab Starting From C1D15 | Arm A Exp Avelumab Starting From C3D1 | Arm B Exp Avelumab Starting From C1D15 | Arm B Exp Avelumab Starting From C3D1 | Arm C Escalation Avelumab Starting From C1D1 | Arm C Exp Avelumab Starting From C1D15 | Arm C Exp Avelumab Starting From C3D1 | Arm D Esc Schedule-1 Dose Level 1; XRT: Starting C1D2 to C1D11 | Arm D Esc Schedule-2 Dose Level 1; XRT: Starting Days -14 to -1 | Arm D Esc Schedule-3 Dose Level 1; XRT: Starting C1D1 to C1D3 | Arm E Esc Schedule-1 Dose Level 1; XRT: Starting C1D2 to C1D11 | Arm E Esc Schedule-2 Dose Level 1; XRT: Starting Days -14 to -1 | Arm F Esc Schedule-1 Dose Level 1; Avelumab Starting From C1D1, XRT: Starting C1D2 to C1D11 | Arm F Esc Schedule-2 Dose Level 1; Avelumab Starting From C1D15, XRT: Starting Days -14 to -1
Number analyzed (Participants) | 13 | 8 | 14 | 10 | 3 | 14 | 9 | 4 | 1 | 7 | 3 | 2 | 4 | 1
Participants | 0 | 3 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Clinical Benefit Rate Per irRECIST
Description: Per irRECIST using CT, MRI,or PET-CT scan: irCR,Disappearance of all target lesions; irPR, >=30% decrease in the sum of the longest diameter of target and new lesions; Immune-related Progressive Disease (irPD), Increase ≥20% of the sum of longest diameter of target and new lesion compared with nadir (minimum 5 mm) or progression of non-target lesions ; Immune-related Stable Disease (irSD), Neither irPR nor irPD; Clinical benefit (CB) = irCR + irPR + irSD ≥6 months.
Time Frame: as for outcome 2
Population: All enrolled patients who were eligible, had received at least one cycle of therapy, and had baseline assessments and at least 1 on-study tumor assessment were considered evaluable for response. Patients who were treated and removed from study prior to on-study tumor assessment because of disease progression were also considered evaluable . In XRT arms, patients were considered evaluable on the study if patients received 75% of radiation dose
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A Exp Avelumab Starting From C1D15 | Arm A Exp Avelumab Starting From C3D1 | Arm B Exp Avelumab Starting From C1D15 | Arm B Exp Avelumab Starting From C3D1 | Arm C Escalation Avelumab Starting From C1D1 | Arm C Exp Avelumab Starting From C1D15 | Arm C Exp Avelumab Starting From C3D1 | Arm D Esc Schedule-1 Dose Level 1; XRT: Starting C1D2 to C1D11 | Arm D Esc Schedule-2 Dose Level 1; XRT: Starting Days -14 to -1 | Arm D Esc Schedule-3 Dose Level 1; XRT: Starting C1D1 to C1D3 | Arm E Esc Schedule-1 Dose Level 1; XRT: Starting C1D2 to C1D11 | Arm E Esc Schedule-2 Dose Level 1; XRT: Starting Days -14 to -1 | Arm F Esc Schedule-1 Dose Level 1; Avelumab Starting From C1D1, XRT: Starting C1D2 to C1D11 | Arm F Esc Schedule-2 Dose Level 1; Avelumab Starting From C1D15, XRT: Starting Days -14 to -1
Number analyzed (Participants) | 13 | 8 | 14 | 10 | 3 | 14 | 9 | 4 | 1 | 7 | 3 | 2 | 4 | 1
Participants | 1 | 3 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0

6. Secondary Outcome: Disease Control Rate Per RECIST v1.1
Description: Per RECIST v1.0 using CT, MRI,or PET-CT scan: CR,Disappearance of all target lesions; PR, >=30% decrease in the sum of the longest diameter of target lesions; PD, Increase ≥20% of the sum of longest diameter compared with nadir (minimum 5 mm) or progression of non-target lesions or new lesion; SD, Neither PR nor PD; Disease control (DC) = CR + PR + SD.
Time Frame: as for outcome 2
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A Exp Avelumab Starting From C1D15 | Arm A Exp Avelumab Starting From C3D1 | Arm B Exp Avelumab Starting From C1D15 | Arm B Exp Avelumab Starting From C3D1 | Arm C Escalation Avelumab Starting From C1D1 | Arm C Exp Avelumab Starting From C1D15 | Arm C Exp Avelumab Starting From C3D1 | Arm D Esc Schedule-1 Dose Level 1; XRT: Starting C1D2 to C1D11 | Arm D Esc Schedule-2 Dose Level 1; XRT: Starting Days -14 to -1 | Arm D Esc Schedule-3 Dose Level 1; XRT: Starting C1D1 to C1D3 | Arm E Esc Schedule-1 Dose Level 1; XRT: Starting C1D2 to C1D11 | Arm E Esc Schedule-2 Dose Level 1; XRT: Starting Days -14 to -1 | Arm F Esc Schedule-1 Dose Level 1; Avelumab Starting From C1D1, XRT: Starting C1D2 to C1D11 | Arm F Esc Schedule-2 Dose Level 1; Avelumab Starting From C1D15, XRT: Starting Days -14 to -1
Number analyzed (Participants) | 13 | 8 | 14 | 10 | 3 | 14 | 9 | 4 | 1 | 7 | 3 | 2 | 4 | 1
Participants | 4 | 7 | 2 | 5 | 1 | 4 | 5 | 2 | 0 | 1 | 1 | 2 | 2 | 0

7. Secondary Outcome: Disease Control Rate Per irRECIST
Description: Per irRECIST using CT, MRI,or PET-CT scan: irCR,Disappearance of all target lesions; irPR, >=30% decrease in the sum of the longest diameter of target and new lesions; irPD, Increase ≥20% of the sum of longest diameter of target and new lesion compared with nadir (minimum 5 mm) or progression of non-target lesions ; irSD, Neither irPR nor irPD; Disease control (DC) = irCR + irPR + irSD.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A Exp Avelumab Starting From C1D15 | Arm A Exp Avelumab Starting From C3D1 | Arm B Exp Avelumab Starting From C1D15 | Arm B Exp Avelumab Starting From C3D1 | Arm C Escalation Avelumab Starting From C1D1 | Arm C Exp Avelumab Starting From C1D15 | Arm C Exp Avelumab Starting From C3D1 | Arm D Esc Schedule-1 Dose Level 1; XRT: Starting C1D2 to C1D11 | Arm D Esc Schedule-2 Dose Level 1; XRT: Starting Days -14 to -1 | Arm D Esc Schedule-3 Dose Level 1; XRT: Starting C1D1 to C1D3 | Arm E Esc Schedule-1 Dose Level 1; XRT: Starting C1D2 to C1D11 | Arm E Esc Schedule-2 Dose Level 1; XRT: Starting Days -14 to -1 | Arm F Esc Schedule-1 Dose Level 1; Avelumab Starting From C1D1, XRT: Starting C1D2 to C1D11 | Arm F Esc Schedule-2 Dose Level 1; Avelumab Starting From C1D15, XRT: Starting Days -14 to -1
Number analyzed (Participants) | 13 | 8 | 14 | 10 | 3 | 14 | 9 | 4 | 1 | 7 | 3 | 2 | 4 | 1
Participants | 7 | 6 | 5 | 5 | 1 | 5 | 5 | 2 | 0 | 2 | 1 | 2 | 2 | 0

ADVERSE EVENTS:
Time Frame: First day of administration of study medication through 30 calendar days after the last administration of the investigational product, through the end of the study up to 3 years.
Description: All AEs were reported regardless of treatment group or relationship to the investigational product(s). AEs were graded per NCI CTCAE v4.03. Every attempt was made to report all SAEs, expected or unexpected, to the IND Office, regardless of attribution within 5 working days and all life-threatening or fatal events, that were unexpected, and related to the study drug within 24 hours (next working day) of knowledge of the event to the Safety Project Manager in the IND Office
Arm/Group | Arm A Exp Avelumab Starting From C1D15 | Arm A Exp Avelumab Starting From C3D1 | Arm B Exp Avelumab Starting From C1D15 | Arm B Exp Avelumab Starting From C3D1 | Arm C Escalation Avelumab Starting From C1D1 | Arm C Exp Avelumab Starting From C1D15 | Arm C Exp Avelumab Starting From C3D1 | Arm D Esc Schedule-1 Dose Level 1; XRT: Starting C1D2 to C1D11 | Arm D Esc Schedule-2 Dose Level 1; XRT: Starting Days -14 to -1 | Arm D Esc Schedule-3 Dose Level 1; XRT: Starting C1D1 to C1D3 | Arm E Esc Schedule-1 Dose Level 1; XRT: Starting C1D2 to C1D11 | Arm E Esc Schedule-2 Dose Level 1; XRT: Starting Days -14 to -1 | Arm F Esc Schedule-1 Dose Level 1; Avelumab Starting From C1D1, XRT: Starting C1D2 to C1D11 | Arm F Esc Schedule-2 Dose Level 1; Avelumab Starting From C1D15, XRT: Starting Days -14 to -1
All-Cause Mortality (participants affected / at risk) | 15/16 | 6/8 | 13/16 | 10/12 | 3/4 | 15/17 | 9/11 | 4/4 | 3/3 | 7/7 | 3/3 | 3/3 | 4/4 | 3/3
Serious Adverse Events (participants affected / at risk) | 8/16 | 6/8 | 3/16 | 7/12 | 3/4 | 6/17 | 5/11 | 4/4 | 3/3 | 0/7 | 1/3 | 1/3 | 4/4 | 2/3
Other Adverse Events (participants affected / at risk) | 15/16 | 8/8 | 14/16 | 11/12 | 4/4 | 15/17 | 11/11 | 4/4 | 2/3 | 7/7 | 3/3 | 3/3 | 4/4 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A Exp Avelumab Starting From C1D15 (N=16) | Arm A Exp Avelumab Starting From C3D1 (N=8) | Arm B Exp Avelumab Starting From C1D15 (N=16) | Arm B Exp Avelumab Starting From C3D1 (N=12) | Arm C Escalation Avelumab Starting From C1D1 (N=4) | Arm C Exp Avelumab Starting From C1D15 (N=17) | Arm C Exp Avelumab Starting From C3D1 (N=11) | Arm D Esc Schedule-1 Dose Level 1; XRT: Starting C1D2 to C1D11 (N=4) | Arm D Esc Schedule-2 Dose Level 1; XRT: Starting Days -14 to -1 (N=3) | Arm D Esc Schedule-3 Dose Level 1; XRT: Starting C1D1 to C1D3 (N=7) | Arm E Esc Schedule-1 Dose Level 1; XRT: Starting C1D2 to C1D11 (N=3) | Arm E Esc Schedule-2 Dose Level 1; XRT: Starting Days -14 to -1 (N=3) | Arm F Esc Schedule-1 Dose Level 1; Avelumab Starting From C1D1, XRT: Starting C1D2 to C1D11 (N=4) | Arm F Esc Schedule-2 Dose Level 1; Avelumab Starting From C1D15, XRT: Starting Days -14 to -1 (N=3)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Autoimmune disorder, hepatitis (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Biliary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Colonic obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Death NOS (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Edema limbs (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Encephalomyelitis infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Endocarditis infective (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Esophageal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Female genital tract fistula (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fever (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal disorders - Gastric outlet obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic Failure (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other, specify (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peritoneal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prolapse of intestinal stoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Serum amylase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thromboembolic event (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tracheostomy site bleeding (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A Exp Avelumab Starting From C1D15 (N=16) | Arm A Exp Avelumab Starting From C3D1 (N=8) | Arm B Exp Avelumab Starting From C1D15 (N=16) | Arm B Exp Avelumab Starting From C3D1 (N=12) | Arm C Escalation Avelumab Starting From C1D1 (N=4) | Arm C Exp Avelumab Starting From C1D15 (N=17) | Arm C Exp Avelumab Starting From C3D1 (N=11) | Arm D Esc Schedule-1 Dose Level 1; XRT: Starting C1D2 to C1D11 (N=4) | Arm D Esc Schedule-2 Dose Level 1; XRT: Starting Days -14 to -1 (N=3) | Arm D Esc Schedule-3 Dose Level 1; XRT: Starting C1D1 to C1D3 (N=7) | Arm E Esc Schedule-1 Dose Level 1; XRT: Starting C1D2 to C1D11 (N=3) | Arm E Esc Schedule-2 Dose Level 1; XRT: Starting Days -14 to -1 (N=3) | Arm F Esc Schedule-1 Dose Level 1; Avelumab Starting From C1D1, XRT: Starting C1D2 to C1D11 (N=4) | Arm F Esc Schedule-2 Dose Level 1; Avelumab Starting From C1D15, XRT: Starting Days -14 to -1 (N=3)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 3 (3) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 4 (4) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Alkaline phosphatase increased (Investigations) | 5 (5) | 5 (5) | 2 (2) | 4 (4) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 3 (3)
Allergic reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Amnesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 5 (5) | 6 (6) | 2 (2) | 3 (3) | 1 (1) | 5 (5) | 4 (4) | 3 (3) | 1 (1) | 2 (2) | 1 (1) | 3 (3) | 1 (1) | 3 (3)
Anorexia (Metabolism and nutrition disorders) | 7 (7) | 1 (1) | 4 (4) | 3 (3) | 1 (1) | 0 (0) | 5 (5) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 5 (5) | 5 (5) | 3 (3) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 3 (3) | 0 (0) | 4 (4) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bile duct stenosis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 5 (5) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac disorders - Other, (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac troponin I increased (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (1)
Cholesterol high (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 5 (5) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CPK increased (Investigations) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Creatinine increased (Investigations) | 2 (2) | 6 (6) | 2 (2) | 0 (0) | 0 (0) | 3 (3) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Death NOS (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Deep vein thrombosis (left leg) (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 2 (2) | 3 (3) | 2 (2) | 3 (3) | 6 (6) | 4 (4) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Edema limbs (General disorders) | 6 (6) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Endocrine disorders - Other, specify (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
epigastric pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye disorders - Other, specify (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 5 (5) | 3 (3) | 3 (3) | 3 (3) | 3 (3) | 3 (3) | 2 (2) | 0 (0) | 2 (2) | 3 (3) | 2 (2) | 2 (2) | 0 (0) | 1 (1)
Fecal incontinence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fever (General disorders) | 3 (3) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flu like symptoms (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroparesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
General disorders and administration site conditions - Other, specify (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hallucinations (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hot flashes (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 2 (2) | 3 (3) | 2 (2) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperphosphatemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
hyperthyroidism (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 4 (4) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 3 (3) | 4 (4) | 0 (0) | 3 (3) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other, specify (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (General disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INR increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Investigations - Other, specify (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 1 (1) | 8 (8) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Lymphedema (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 4 (4) | 3 (3) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatic enzymes decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paresthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Photosensitivity (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Psychiatric disorders - Adjustment disorder with depressive mood (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Rash pustular (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal fistula (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Reproductive system and breast disorders - Other, specify (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Serum amylase increased (Investigations) | 2 (2) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sprain: left ankle (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Swelling: left ankle (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Testicular pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thromboembolic event (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal hemorrhage (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vaginal inflammation (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Weight loss (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cell decreased (Investigations) | 3 (3) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-24): https://cdn.clinicaltrials.gov/large-docs/47/NCT03217747/Prot_SAP_000.pdf